CLINICAL TRIAL: NCT06516731
Title: A Single Group Study to Evaluate the Effects of a pH Balanced Cleanser on Women's Intimate Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Love Wellness (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20401
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Vaginal Health; Vaginal pH
Keywords: pH Balanced Cleanser; Vaginal Health; Women's Health; Intimate Hygiene; Intimate Skin Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pH Balanced Cleanser (Experimental): Participants will use the pH Balanced Cleanser daily during showers. The study will evaluate the effects on vulvar and vaginal health, including odor and pH levels, and assess the tolerability of the product.
  Interventions: Dietary Supplement: pH Balanced Cleanser

INTERVENTIONS:
Dietary Supplement: pH Balanced Cleanser — Participants will use the pH Balanced Cleanser daily during showers. The cleanser should be applied to the vulva with clean hands, gently worked into a lather, and rinsed clean. Participants will complete baseline and weekly questionnaires and vaginal pH tests over an 8-week period to evaluate the effects on vulvar and vaginal health, including odor and pH levels, and assess the tolerability of the product.
  Other Names: Love Wellness pH Balanced Cleanser

SUMMARY:
This virtual single-group study will last 8 weeks, involving the daily use of a pH Balanced Cleanser by 40 female participants. The study aims to evaluate the effect of the cleanser on signs of vulvar and vaginal health and its tolerability.

DETAILED DESCRIPTION:
Participants will use the Love Wellness pH Balanced Cleanser daily during showers. Questionnaires will be completed at Baseline, first use, Week 2, Week 4, Week 6, and Week 8. Vaginal pH testing will be conducted weekly using Vaginox vaginal pH testing strips. The primary objective is to assess parameters of vulvar and vaginal health, while the secondary objective is to evaluate product tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18+
* Self-reported issues with vaginal odor, itching, or intimate skin discomfort
* Previous use of vaginal cleansers without severe adverse reactions
* Generally healthy without uncontrolled chronic diseases
* Willing to avoid intra-vaginal products during the study
* Consistent use of any vaginal health-targeted supplements for at least 3 months prior

Exclusion Criteria:

* Pre-existing chronic conditions preventing protocol adherence
* Planned reproductive health procedures
* Recent changes in medications or supplements targeting vaginal health
* Known severe allergic reactions
* Pregnancy, breastfeeding, or attempting to conceive
* Unwillingness to follow study protocol
* History of vaginal, cervical, vulvar, uterine, or ovarian cancer
* Recent changes or discontinuation of hormonal birth control
* Recent surgeries or invasive treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Effect of pH Balanced Cleanser on Vulvar and Vaginal Health | Baseline, first use, Week 2, Week 4, Week 6, Week 8
  Parameters associated with vulvar and vaginal health, including odor and pH levels, will be evaluated. Participants will complete questionnaires at Baseline, first use, Week 2, Week 4, Week 6, and Week 8.
Effect of pH Balanced Cleanser on Vulvar and Vaginal Health | Baseline and Week 8
  Vaginal pH testing will be conducted weekly from Baseline to Week 8.

SECONDARY OUTCOMES:
Tolerability of pH Balanced Cleanser | Baseline, first use, Week 2, Week 4, Week 6, Week 8
  The tolerability of the product will be evaluated via questionnaires at first use, Week 2, Week 4, Week 6, and Week 8. Parameters of interest include reported irritation or itchiness associated with the product, comfort when using the product, negative changes in vaginal pH associated with product use, and participants' overall perceptions of the product.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No